CLINICAL TRIAL: NCT04840667
Title: A Phase 3, Open-label Study to Evaluate the Efficacy and Safety of REPLAGAL® in Treatment-naïve Subjects With Fabry Disease
Brief Title: A Study of Replagal in Treatment-naïve Adults With Fabry Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study closed due to enrolment challenges, not for any safety issues
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP675-301; 2018-004689-32 (EudraCT Number)
Record Dates: First submitted 2020-07-07; First posted 2021-04-12 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REPLAGAL (Experimental): Participants will receive REPLAGAL 0.2 milligram per kilogram (mg/kg) body weight of intravenous (IV) infusion Every Other Week (EOW) for 104 weeks.
  Interventions: Drug: REPLAGAL

INTERVENTIONS:
Drug: REPLAGAL — Participants will receive REPLAGAL 0.2 mg/kg body weight of IV infusion for 104 weeks.
  Other Names: SHP675

SUMMARY:
In this study, adults with Fabry Disease who have not had any treatment for this condition will be treated with Replagal. The main aim of the study is to check if Replagal improves kidney function and heart structure of participants with Fabry Disease. Participants will receive one Replagal infusion every other week for up to 104 weeks. They will visit the clinic every 12 to 14 weeks during treatment with a follow-up visit 2 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participant must voluntarily sign an Institutional Review Board (IRB)/Independent Ethics Committee/Research Ethics Board approved informed consent form after all relevant aspects of the study have been explained and discussed with the participant.
* The participant has Fabry disease as confirmed at screening by the following criteria using a dried blood spot (DBS) assay:

  1. For male participants, Fabry disease is confirmed by a deficiency of alpha-galactosidase A (GLA) activity and a mutation in the GLA gene
  2. For female participants, Fabry disease is confirmed by a mutation in the GLA gene
* The participant is 18 to 65 years of age, inclusive.
* Female participants must have a negative pregnancy test at screening.
* Female participants of child-bearing potential must agree to use a medically acceptable method of contraception at all times during the study and for at least 14 days after the final study infusion; the methods of acceptable contraception are listed in the protocol.
* The participant is deemed, as determined by the investigator, to have adequate general health to undergo the specified protocol-related procedures and to have no safety or medical contraindications for participation.
* The participant has not received any treatment (approved or investigational) specific to Fabry disease, such as enzyme replacement therapy (ERT), chaperone therapy, or substrate reduction therapy.
* The participant must have an eGFR of 45 to 120 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2); eGFR will be calculated by a Shire-designated laboratory using the CKD-EPI formula. If the eGFR measurement at screening is not within the range, a second eGFR measurement may be completed and, if in range, used as the screening value. If a second measurement is taken, a minimum of 1 week and maximum of 30 days should separate it from the first. This inclusion criterion follows the European Guidelines for Treatment of Fabry Disease and Kidney Disease Improving Global Outcomes guidelines for classification of renal disease.
* The participant has left ventricular hypertrophy (LVH), where LVH is defined as left ventricular mass index (LVMI) greater than (>) 50 gram per square meter (g/m^2.7) confirmed by cardiac magnetic resonance imaging (cMRI) at screening. The cMRI value at screening will serve as the baseline value.

Exclusion Criteria:

* In the opinion of the investigator, the participant's life expectancy is less than or equal to (<=) 5 years.
* The participant has undergone or is scheduled to undergo kidney transplantation or is currently on dialysis, or has any signs or symptoms of end stage renal disease.
* Urine protein/creatinine ratio (PCR) greater than (>) 1.5 milligram per milligram (mg/mg).
* Participants who have clinically relevant history of allergy or signs or symptoms of severe hypersensitivity, (including hypersensitivity to the REPLAGAL active substance or any of the excipients), which in the investigator's judgment, will substantially increase the participant's risk if he or she participates in the study.
* Cardiac fibrosis involving more than 2 segments, as determined by cMRI at screening.
* In the opinion of the investigator, the participant has non-Fabry disease-related cause of end-organ (renal, cardiac, central nervous system) dysfunction/failure or is receiving medications that may affect the rate of disease progression, as assessed by cardiac and/or renal measures.
* The participant has a positive test at screening for hepatitis B surface antigen, positive test for hepatitis B core antibody, positive test for hepatitis C (HCV) antibody with confirmation by HCV-ribonucleic acid polymerase chain reaction testing, or positive test for human immunodeficiency virus antibody.
* Treatment with REPLAGAL at any time prior to the study.
* Prior treatment with any of the following medications:

  1. FABRAZYME (agalsidase beta) and its biosimilars
  2. GLYSET (miglitol)
  3. ZAVESCA (miglustat)
  4. CERDELGA (eliglustat)
  5. GALAFOLD (migalastat)
  6. Any investigational product for treatment of Fabry disease
* Treatment at any time during the study with the following medications:

  1. Chloroquine
  2. Amiodarone
  3. Monobenzone
  4. Gentamicin
* The participant is pregnant or lactating.
* The participant has a body mass index > 39 kilogram per square meter (kg/ m^2). (Body mass index [BMI] = kg/ m^2).
* The participant is treated or has been treated with any investigational drug within 30 days of study start.
* The participant is unable to understand the nature, scope, and possible consequences of the study.
* The participant is unable to comply with the protocol, eg, uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for evaluations, or is otherwise unlikely to complete the study, as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (28):
- Canada (2):
  - M.A.G.I.C. Clinic Ltd. Metabolics and Genetics in Calgary, Calgary
  - Queen Elizabeth II Health Sciences Center, Halifax
- Finland (2):
  - Turun Yliopistollinen Keskussairaala, Turku
  - Vaasan Keskussairaala, Vaasa
- Germany (5):
  - Charité - Universitätsklinikum, Berlin
  - SphinCS, Höchheim
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Fachinternistische Gemeinschaftspraxis, Müllheim
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (6):
  - Laiko General Hospital of Athens, Athens
  - Attikon University General Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - Onasseio Private Practise Hospital of Piraeus, Kallithea
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Poland (3):
  - Szpital Uniwersytecki, Krakow
  - Narodowy Instytut Kardiologii im Prymasa Tysiaclecia Kardynala Stefana Wyszynskiego - Instytut Badaw, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Portugal (3):
  - Centro Hospitalar e Universitário de Coimbra EPE, Coimbra
  - Hospital Senhora da Oliveira - Guimaraes, E.P.E, Guimarães
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
- Spain (6):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de Torrecárdenas, Almería
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Quironsalud Zaragoza, Zaragoza
- Akademiska Sjukhuset I Uppsala, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
The study was terminated by the Sponsor due to enrolment challenges. No participants were evaluated, and no data were collected.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61147ce4cd353f0032b92064

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 17 participants were screened and signed informed consent but none of the participants received any treatment due to screen failures. The study was terminated by the sponsor due to enrolment challenges and no participants were treated, therefore no data were evaluated and collected to be reported in this study.
Groups:
- REPLAGAL: Participants were to receive REPLAGAL 0.2 milligram per kilogram (mg/kg) body weight of intravenous (IV) infusion every other week (EOW) for 104 weeks.
Period: Overall Study
Arm/Group | REPLAGAL
Started | 17
Treated | 0
Completed | 0
Not Completed | 17
Not completed — Screen failures/ Failure to meet inclusion criteria | 17

BASELINE CHARACTERISTICS:
Population: A total of 17 participants were screened and signed informed consent but none of the participants received any treatment due to screen failures. The study was terminated by the sponsor due to enrolment challenges and no participants were treated, therefore no data were evaluated and collected to be reported in this study.
Groups:
- REPLAGAL: Participants were to receive REPLAGAL 0.2 mg/kg body weight of IV infusion EOW for 104 weeks.
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Race/Ethnicity, Customized

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Renal Function at Week 104
Description: Renal function was planned to be assessed by estimated glomerular filtration rate (eGFR) using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. The eGFR was planned to be calculated by CKD-EPI formula: eGFR = 141 x min (Serum Creatinine [Scr]/κ,1)^(α) x max(Scr/κ,1)^(-1.209) x 0.993^(Age) x 1.018 (if female) x 1.159 (if black) where: Scr was serum creatinine (mg/dL); κ was 0.7 for females and 0.9 for males; α was -0.329 for females and -0.411 for males; min indicated the minimum of Scr/κ or 1; max indicated the maximum of Scr /κ or 1. Change from baseline in renal function at Week 104 was planned to be reported.
Time Frame: Baseline, Week 104
Population: The study was terminated by the Sponsor due to enrolment challenges. No participants were treated in this study, therefore no data were evaluated and collected for this outcome measure.
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline in Cardiac Structure at Week 104
Description: Cardiac structure was planned to be assessed by left ventricular mass index (LVMI) using cardiac magnetic resonance imaging (cMRI). Change from baseline in cardiac structure at Week 104 was planned to be reported.
Time Frame: Baseline, Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

3. Secondary Outcome: Annualized Rate of Change in Estimated Glomerular Filtration Rate (eGFR) up to Week 104
Description: Annualized rate of change in eGFR up to Week 104 was planned to be reported.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

4. Secondary Outcome: Annualized Rate of Change in Left Ventricular Mass Index (LVMI) up to Week 104
Description: Annualized rate of change in LVMI up to Week 104 was planned to be reported.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in eGFR up to Week 104
Description: Change from baseline in eGFR up to Week 104 was planned to be reported.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in LVMI up to Week 104
Description: Change from baseline in LVMI up to Week 104 was planned to be reported.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Proteinuria up to Week 104
Description: Proteinuria was to be measured based on protein/creatinine ratio (PCR). Change from baseline in proteinuria up to Week 104 was planned to be reported.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Cardiac Fibrotic Segments up to Week 104
Description: Change from baseline in cardiac fibrotic segments suggestive of cardiac fibrosis up to Week 104 was planned to be assessed by volume of fibrosis, measured by cMRI.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Interventricular Septal End-Diastolic Thickness and Posterior Wall Thickness in Diastole up to Week 104
Description: Change from baseline in interventricular septal end-diastolic thickness and posterior wall thickness in diastole up to Week 104 was planned to be measured by cMRI.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Plasma Globotriaosylsphingosine (Lyso-Gb3) up to Week 104
Description: Change from baseline in lyso-Gb3 up to Week 104 was planned to be reported.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Time Frame: From start of study drug administration up to follow-up visit (i.e., up to Week 106)
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants Who Will Develop Anti-drug Antibodies (ADA) to REPLAGAL
Description: Number of participants who will develop ADA to REPLAGAL was planned to be reported.
Time Frame: From Baseline up to Week 104
Population: as for outcome 1
Arm/Group | REPLAGAL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected in this study
Description: The study was terminated by the Sponsor due to enrolment challenges. No participants were treated, therefore no Death, SAE and NSAEs data were evaluated and collected to be reported in this study.
Arm/Group | REPLAGAL
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor due to enrolment challenges. No participants were evaluated, and no data were collected to be reported in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT04840667/Prot_SAP_000.pdf